CLINICAL TRIAL: NCT03493568
Title: Open Label, Randomized (1:1) Clinical Trial to Evaluate Switching From Dual Regimens Based on Dolutegravir Plus a Reverse Transcriptase Inhibitor to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed, HIV-1 Infected Patients (Be-OnE Study).
Brief Title: Switch From Dual Regimens Based on Dolutegravir Plus a Reverse Transcriptase Inhibitor to E/C/F/TAF in Virologically Suppressed, HIV-1 Infected Patients (Be-OnE)
Acronym: Be-OnE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The futility analysis on 24-week results estimated that there was only 2% probability of verifying the study hypothesis of a higher proportion pat. with no residual viremia through 48w in arm E/C/F/TAF
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Castagna Antonella, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Be-OnE Study
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; dolutegravir

STUDY DESIGN:
Intervention Model Description: Treatments
  1. Genvoya 150Mg-150Mg-200Mg-10Mg Tablet ( 1 pill every 24 hours)
  2. Dolutegravir 50 mg (1 pill every 24 hours) plus one Reverse Trascriptase Inhibitor (at label dose)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genvoya 150Mg-150Mg-200Mg-10Mg Table (Experimental): switch to the treatment Genvoya 150Mg-150Mg-200Mg-10Mg Table (1 pill every 24 hour)
  Interventions: Drug: Genvoya 150Mg-150Mg-200Mg-10Mg Tablet
- Dolutegravir 50 mg plus one RTI (at label dose) (Active Comparator): Continuing Dolutegravir 50 mg (1 pill every 24 hours) plus one RTI (at label dose)
  Interventions: Drug: Dolutegravir 50 mg plus one RTI

INTERVENTIONS:
Drug: Genvoya 150Mg-150Mg-200Mg-10Mg Tablet — switch to Genvoya 150Mg-150Mg-200Mg-10Mg Tablet in patients virologically suppressed HIV-1 infected patients.
  Arms: Genvoya 150Mg-150Mg-200Mg-10Mg Table
Drug: Dolutegravir 50 mg plus one RTI — Continuing Dolutegravir 50 mg (1 pill every 24 hours) plus one RTI (at label dose)
  Arms: Dolutegravir 50 mg plus one RTI (at label dose)

SUMMARY:
Research hypothesis:

Switching from dual regimens based on dolutegravir plus a RTI to a single tablet regimen of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF), lowers the exposure to Residual Viremia (and hence the risk of viral rebound), without increasing treatment toxicity.

DETAILED DESCRIPTION:
Study design Randomized, single-center, open-label, 96-week superiority study. Patients with HIV-RNA <50 copies/mL while receiving DTG plus one RTI will be randomized 1:1 to continue the ongoing treatment or to switch to E/C/F/TAF.

Randomization list will be a computer-generated list (with equal block sizes) and will be incorporated within an electronic clinical report form (eCRF).

Patients will be evaluated at screening, baseline, week 4, 8, 16, 24, 32, 40, 48, 60, 72, 84, 96 or premature discontinuation.

At each visit the following evaluations will be performed:

1. clinical assessment.
2. routine laboratory tests (hematological tests and clinical chemistry). Additional blood samples will be collected at specified visits for storage and further determinations (e.g. RV by a single-copy assay).

During follow-up, at different timepoints, patients will additionally undergo HIV-DNA quantification in PBMCs (BL, 48 and 96 weeks) and quality of life (QOL) and adherence assessement (BL, 48 and 96 weeks).

Viral load will be assessed by Abbott Real time PCR (Abbott RealTime HIV-1) Residual viremia (RV) will be defined as any detectable HIV-RNA value below 50 copies/mL Virologic failure will be defined as a confirmed rebound in plasma HIV-RNA levels ≥ 50 copies/mL

Subjects who meet a protocol-defined virologic failure during follow-up will be discontinued from the study.

At virologic failure subjects will perform genotypic HIV resistance testing and a determination in plasma of elvitegravir or DTG Cthrough.

HIV-DNA will be extracted from 1x106 peripheral blood mononuclear cells (PBMCs) by using Qiagen DNA extraction kit and quantified by Real Time PCR (ABI Prism 7900).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Willing and able to provide informed consent
3. On a stable (at least 3 months) antiretroviral therapy with DTG 50 mg QD plus one RTI
4. HIV-RNA <50 copies/mL since at least 6 months

Exclusion Criteria:

1. Active AIDS-defining condition (except Kaposi's sarcoma non requiring systemic chemotherapy)
2. Serious illness requiring systemic treatment and/or hospitalization
3. Current use of immunomodulant or immunosuppressive drugs
4. Need (or will likely need) of treatment with antacids
5. Use of drugs contraindicated with study drugs, according to technical sheets
6. Previous suboptimal therapies with NRTIs or presence of TAMs (type 1 or 2) in previous resistance tests (patients with the 184I/V mutation alone are allowed to enter the study)
7. Resistance or previous virological failure to InSTIs
8. Detectable HCV-RNA
9. Documented allergy to COBI or EVG or FTC or tenofovir.
10. Absolute neutrophil count (ANC) <500/µL
11. Haemoglobin <8.0 g/dL
12. Platelet count <50,000/µL
13. eGFR <30 mL/min/1.73m2 by CKD-EPI equation
14. Alanine aminotransferase (ALT) more than 5 times the upper limit of normal (ULN)
15. Presence of Child Pugh Class B or C liver cirrhosis.
16. Pregnancy or breastfeeding
17. Woman of childbearing potential who does not agree to adopt highly effective contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Residual Viremia | 48 weeks
  To investigate RV through 48 weeks in virologically suppressed patients randomized to continue treatment with DTG plus a single RTI or to switch to E/C/F/TAF.

SECONDARY OUTCOMES:
virological rebound | 48 weeks
  To investigate the occurrence of virological rebound above 50 HIV-RNA copies/mL;
viral reservoir | 48 weeks
  To investigate changes in viral reservoir (HIV-DNA)
QOL | 48 weeks
  To investigate changes in the quality of life (administration of questionnaire ISSQoL uses five- point Likert scales 1 never 2 rarely 3 sometimes 4 often 5 always)
Adherence | 48 weeks
  To investigate changes in adherence (administration of questionnaire uses scale ranges from 0 to 100)
Virological failure | 96 weeks
  proportion of patient in virological rebound
viral reservoir | 96 weeks
  change in viral reservoir (HIV-DNA extracted from peripheral blood mononuclear cells by using Qiagen DNA extraction kit and quantified by Real Time PCR)
QOL | 96 weeks
  To investigate changes in the quality of life (administration of questionnaire To investigate changes in the quality of life (administration of questionnaire ISSQoL uses five- point Likert scales 1 never 2 rarely 3 sometimes 4 often 5 always))
Adherence. | 96 weeks
  To investigate changes in adherence (administration of questionnaire uses scale ranges from 0 to 100 )

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Lazzarin, Prof, Principal Investigator — Ospedale San Raffaele
Locations (2):
- Italy (2):
  - Ospedale San Raffaele, Milan, Lombardy
  - Ospedale San Raffaele Scientific Institute, Milan

IPD SHARING:
Plan to Share IPD: Yes
Data shared in Scientific Congress (abstract and pubblications)

REFERENCES:
- [Background] Margolis DA, Brinson CC, Smith GHR, de Vente J, Hagins DP, Eron JJ, Griffith SK, Clair MHS, Stevens MC, Williams PE, Ford SL, Stancil BS, Bomar MM, Hudson KJ, Smith KY, Spreen WR; LAI116482 Study Team. Cabotegravir plus rilpivirine, once a day, after induction with cabotegravir plus nucleoside reverse transcriptase inhibitors in antiretroviral-naive adults with HIV-1 infection (LATTE): a randomised, phase 2b, dose-ranging trial. Lancet Infect Dis. 2015 Oct;15(10):1145-1155. doi: 10.1016/S1473-3099(15)00152-8. Epub 2015 Jul 19. PMID 26201299
- [Background] Riddler SA, Aga E, Bosch RJ, Bastow B, Bedison M, Vagratian D, Vaida F, Eron JJ, Gandhi RT, Mellors JW; ACTG A5276s Protocol Team. Continued Slow Decay of the Residual Plasma Viremia Level in HIV-1-Infected Adults Receiving Long-term Antiretroviral Therapy. J Infect Dis. 2016 Feb 15;213(4):556-60. doi: 10.1093/infdis/jiv433. Epub 2015 Sep 2. PMID 26333941
- [Background] Gianotti N, Canducci F, Galli L, Cossarini F, Salpietro S, Poli A, Nozza S, Spagnuolo V, Clementi M, Sampaolo M, Ceresola ER, Racca S, Lazzarin A, Castagna A. HIV DNA loads, plasma residual viraemia and risk of virological rebound in heavily treated, virologically suppressed HIV-infected patients. Clin Microbiol Infect. 2015 Jan;21(1):103.e7-103.e10. doi: 10.1016/j.cmi.2014.08.004. Epub 2014 Oct 13. PMID 25636935
- [Background] Gianotti N, Galli L, Salpietro S, Cernuschi M, Bossolasco S, Maillard M, Spagnuolo V, Canducci F, Clementi M, Lazzarin A, Castagna A. Virological rebound in human immunodeficiency virus-infected patients with or without residual viraemia: results from an extended follow-up. Clin Microbiol Infect. 2013 Dec;19(12):E542-4. doi: 10.1111/1469-0691.12266. Epub 2013 Jul 24. PMID 23890370
- [Background] Maggiolo F, Callegaro A, Cologni G, Bernardini C, Velenti D, Gregis G, Quinzan G, Soavi L, Iannotti N, Malfatto E, Leone S. Ultrasensitive assessment of residual low-level HIV viremia in HAART-treated patients and risk of virological failure. J Acquir Immune Defic Syndr. 2012 Aug 15;60(5):473-82. doi: 10.1097/QAI.0b013e3182567a57. PMID 22481602
- [Background] Doyle T, Smith C, Vitiello P, Cambiano V, Johnson M, Owen A, Phillips AN, Geretti AM. Plasma HIV-1 RNA detection below 50 copies/ml and risk of virologic rebound in patients receiving highly active antiretroviral therapy. Clin Infect Dis. 2012 Mar 1;54(5):724-32. doi: 10.1093/cid/cir936. Epub 2012 Jan 11. PMID 22238167
- [Background] Mills A, Arribas JR, Andrade-Villanueva J, DiPerri G, Van Lunzen J, Koenig E, Elion R, Cavassini M, Madruga JV, Brunetta J, Shamblaw D, DeJesus E, Orkin C, Wohl DA, Brar I, Stephens JL, Girard PM, Huhn G, Plummer A, Liu YP, Cheng AK, McCallister S; GS-US-292-0109 team. Switching from tenofovir disoproxil fumarate to tenofovir alafenamide in antiretroviral regimens for virologically suppressed adults with HIV-1 infection: a randomised, active-controlled, multicentre, open-label, phase 3, non-inferiority study. Lancet Infect Dis. 2016 Jan;16(1):43-52. doi: 10.1016/S1473-3099(15)00348-5. Epub 2015 Nov 2. PMID 26538525
- [Background] Palmer S, Wiegand AP, Maldarelli F, Bazmi H, Mican JM, Polis M, Dewar RL, Planta A, Liu S, Metcalf JA, Mellors JW, Coffin JM. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID 14532178